CLINICAL TRIAL: NCT03898115
Title: Effect of a Multifaceted Implementation Program on Compliance of Daily Chlorohexidine Bathing in Critical Care and Bone Marrow Units
Brief Title: Implementation Program to Improve CHG Bathing Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00101819
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2020-02

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)
Keywords: implementation science; chlorhexidine gluconate bathing

STUDY DESIGN:
Intervention Model Description: This study will be multicenter, cluster randomized, step-wedged design. The unit of randomization will be the inpatient units admitted critically ill patients, with the initial intervention being carried out over 4 months. The study plans to enroll approximately 14 units at 2 sites. Four sequences will be enrolled into the intervention each month; each sequence will have 3-4 units
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHG Bathing Implementation (Experimental): In a step-wedged design, ICUs and BMT units will be enrolled into a educational program to improve knowledge/compliance with daily CHG bathing
  Interventions: Behavioral: CHG Education
- Control (No Intervention): In a step-wedged design, ICUs and BMT units will be enrolled over a rolling 4 month time frame; when not enrolled, this data will serve as control data

INTERVENTIONS:
Behavioral: CHG Education — The CHG educational intervention will include "educational outreach" and "audit and feedback" implementation strategies
  Arms: CHG Bathing Implementation

SUMMARY:
This study will be a multicenter, cluster randomized, step-wedged design. The unit of randomization will be the inpatient units admitted critically ill patients, with the interventions being carried out over 4 months. The study plans to enroll 14 units at 2 sites. Four sequences will be enrolled into the intervention each month; each sequence will have 3-4 units (see figure 1).

Units eligible for the study will have patients that are critically ill admitted and have had at least 1 CLABSI events over the past 12 months (fiscal year). Given the pragmatic nature of the study design, there will be limited additional inclusion and exclusion criteria. Prior to the beginning the study, all nursing staff (RNs and nursing assistants [NAs]) will receive a survey link (RedCAP) to understand their perceptions of CHG bathing. After all units have been enrolled (approximately 4 months), nursing staff will be sent a post-survey to see if their perceptions have improved after the program. Further, the Context Assessment Index (used with permission; via RedCAP) will also be used to assess the context (i.e., culture) in which clinicians works and the effect this has on using evidence in practice. This will be provided to infection prevention champions on each unit one time, at the beginning of enrollment.

All hospitals in the trial will receive access to site-level quality reports on CLABSI data. The interventions will include a "direct engagement" at the site level; this strategy will build upon current quality improvement interventions developed from the Agency for Healthcare Research & Quality for optimization of care for critically ill patients at risk for CLABSIs. The multidisciplinary teams will include national key opinion leaders in quality improvement working with local infection prevention specialists and support staff to help healthcare systems and hospitals design or revise quality improvement plans. Units will receive feedback on quality improvement efforts, including audit and feedback reviewing their CHG bathing compliance and CLABSI rates. Duke will serve as the primary statistical center and analysis will be generated by Duke. The only risk in this study is the possibility of breach of confidentiality.

The primary objective of this study is to assess the effect of a customized, multifaceted quality improvement [QI] program on compliance with daily chlorhexidine gluconate (CHG) bathing per the AHRQ protocol in inpatient units that admit critically ill patients. Further, we will assess the effect of this program on nursing staffs' perception of the importance of CHG bathing. The Context Assessment Index (used with permission) will also be used to assess the context (i.e., culture) in which clinicians works and the effect this has on using evidence in practice. The secondary objective of this study is to examine the effect of the QI program on central line-associated bloodstream infection (CLABSI) rates. Primary outcomes and CLABSI rates will be measured at 12 months to assess sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Units eligible for the study will have patients that are critically ill admitted and have had at least 1 CLABSI events over the past 12 months (fiscal year).

Exclusion Criteria:

* Units with 0 CLABSIs over the past 12 months (fiscal year).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
CHG Bathing Documentation Compliance | Span of 17 months total (initial intervention May - Oct. 2019; sustainability Sept. 2020)
  (1) Compliance of daily CHG bathing documentation (measured via documentation audits)
CHG Bathing Process Compliance | Span of 17 months total (initial intervention May - Oct. 2019; sustainability Sept. 2020)
  (2) Compliance of CHG bathing process (measured via observational audits)

SECONDARY OUTCOMES:
Unit Culture | Pre (month 0); will be open for 2 weeks
  (3) Unit culture (measured via the Context Assessment Index)
Staff perceptions/knowledge of CHG bathing | Pre (month 0) and post (170 weeks later)
  (4) Nursing staffs' perceptions of CHG bathing (measured via a Qualtrics pre- and post-survey of 24 total questions; 12 demographic and 12 related to CHG bathing)
CLABSIs | May 2019 - September 2020 (17 months total)
  (5) CLABSI rates (measured via current National Healthcare Safety Network [NHSN] processes)

CONTACTS AND LOCATIONS:
Overall Officials: Staci Reynolds, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Hospital, Durham, North Carolina
  - Wake Med, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers.

REFERENCES:
- [Background] Reynolds SS, Granger BB, Hatch D. Self-Reported versus observed audit: Measuring CHG bathing compliance. Am J Infect Control. 2021 Dec;49(12):1575-1577. doi: 10.1016/j.ajic.2021.08.019. Epub 2021 Aug 22. PMID 34433015
- [Background] Woltz PC, Granger BB, Reynolds SS. Measuring and Evaluating Clinical Context in Implementation Science Research. AACN Adv Crit Care. 2022 Mar 15;33(1):103-110. doi: 10.4037/aacnacc2022664. No abstract available. PMID 35259215
- [Background] Reynolds SS, Woltz P, Neff J, Elliott J, Granger BB. Impact of an Implementation Science Study on Nursing Leader Competencies: A Qualitative Study. Nurse Leader. 2022; 20(1): 70-74.
- [Result] Reynolds SS, Woltz P, Keating E, Neff J, Elliott J, Hatch D, Yang Q, Granger BB. Results of the CHlorhexidine Gluconate Bathing implementation intervention to improve evidence-based nursing practices for prevention of central line associated bloodstream infections Study (CHanGing BathS): a stepped wedge cluster randomized trial. Implement Sci. 2021 Apr 26;16(1):45. doi: 10.1186/s13012-021-01112-4. PMID 33902653
- [Result] Reynolds SS, Woltz P, Keating E, Neff J, Elliott J, Granger BB. Program Evaluation of Implementation Science Outcomes From an Intervention to Improve Compliance With Chlorhexidine Gluconate Bathing: A Qualitative Study. Dimens Crit Care Nurs. 2022 Jul-Aug 01;41(4):200-208. doi: 10.1097/DCC.0000000000000530. PMID 35617584